CLINICAL TRIAL: NCT04395599
Title: Assessment of Air Contamination Risk by Sars-Cov2 During Visceral Surgery in COVID19 Patients: Pilot Study.
Brief Title: Risk of Air Contamination During Visceral Surgery in COVID19 Patients
Acronym: COELIOCOVID
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Lille (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 2020_44; 2020-A01461-38 (Other: ID-RCB number,ANSM)
Record Dates: First submitted 2020-05-19; First posted 2020-05-20 (Actual); Last update posted 2025-12-23 (Actual); Status verified 2025-12

CONDITIONS: Sars-CoV2; Surgery; COVID
Keywords: COVID-19; visceral surgery; air contamination; laparoscopy, prevention; prevention
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Intervention Model Description: COVID19 patients undergoing visceral surgery
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- COVID19 patients undergoing visceral surgery (Experimental)
  Interventions: Other: Cartography of air contamination, environment contamination and biological fluid by Sars-Cov2 during visceral surgery in COVID19 patients.

INTERVENTIONS:
Other: Cartography of air contamination, environment contamination and biological fluid by Sars-Cov2 during visceral surgery in COVID19 patients. — Air sampling, operating room surfaces sampling and patients' biological fluid sampling for Sars-Cov2 quantification

SUMMARY:
Sars-Cov2 has been found in the digestive tract, as well as the respiratory tract. Protection of health care workers during surgery has been increased and some guidelines advocate for abandoning laparoscopy in COVID19 patients for fear of contamination, evenghtough this does not benefit the patient. However, Sars-Cov2 contamination risk during visceral surgery remains unknown. Inadequate protection is unnecessary costful and can be inefficient if too binding. Our hypotheses are that 1) Sars-Cov 2 can travel through droplet and air during visceral surgery. 2) Laparoscopy, because of the pneumoperitoneum and its leaks, warrant more air contamination whereas laparotomy warrant more droplet contamination, which would justified increased protection.

ELIGIBILITY:
Inclusion Criteria:

* Documented Sars-Cov2 infection (nasopharyngeal swab, tracheal sampling, thoracic CT, serology)
* Need of visceral surgery (laparoscopy or laparotomy)
* Signed informed consent
* Social coverage
* Patient who agrees to be included in the study and who signs the informed consent form
* Patient affiliated to a healthcare insurance plan
* Patient willing to comply with study's requirements

Exclusion Criteria:

* Need of another type of surgery during the same procedure
* Mentally unbalanced patients, under supervision or guardianship
* Patient who does not understand French/ is unable to give consent
* Patient not affiliated to a French or European healthcare insurance
* Patient incarcerated

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2021-11-16 (Actual); Primary Completion 2022-01-27 (Actual); Study Completion 2022-01-27 (Actual)

PRIMARY OUTCOMES:
Air contamination | 10 minutes after incision if no opening of the digestive lumen, or 10 minutes after opening of the digestive tract
  Composite criteria: "50cm above the operating site" and/or "1m50 from the operating site" and/or "3m from the operating site"

SECONDARY OUTCOMES:
Environment contamination | At the end of surgery, an average 1 hour 30 min
  Cartography of Sars-Cov2 environment surface contamination
Surgical approach | At the end of the intervention, an average 2 hours
  Composite criteria: air contamination or environment contamination positivity rate according to surgical approach (laparoscopy or laparotomy)
Opening of the digestive tract | At the end of the intervention,an average 2 hours
  Composite criteria: air contamination or environment contamination positivity rate according to opening of digestive tract status (opened or not)
Biological fluids | During the procedure, an average 2 hours 30 min
  Cartography of Sars-Cov2 presence in biological fluids (blood, stools, peritoneal fluid, digestive fluids, sputum, bile)
Pneumoperitoneum | At the end of the procedure,an average 2 hours 30 min
  Presence of Sars-Cov 2 in pneumoperitoneum, evaluated on surgical smoke filter

CONTACTS AND LOCATIONS:
Overall Officials: Robert CAIAZZO, MD,PhD, Principal Investigator — University Hospital, Lille
Locations (1):
- Hop Claude Huriez Chu Lille, Lille, France

IPD SHARING:
Plan to Share IPD: No